CLINICAL TRIAL: NCT05725252
Title: Phase 1 Study to Evaluate the Safety and the Pharmacokinetics of NVP-2203 in Healthy Adult Volunteers
Brief Title: To Evaluate the Safety and the Pharmacokinetics of NVP-2203
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: NVP Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NVP-2203_BA
Record Dates: First submitted 2023-01-24; First posted 2023-02-13 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2023-10

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NVP-2203 (Experimental): After fasting (except water) for at least 10 hours before dosing, oral administration of investigational product once daily on Period 1(or Period 2)
  Interventions: Drug: NVP-2203
- NVP-2203-R (Active Comparator): After fasting (except water) for at least 10 hours before dosing, oral administration of investigational product once daily on Period 1(or Period 2)
  Interventions: Drug: NVP-2203-R

INTERVENTIONS:
Drug: NVP-2203 — NVP-2203(Combination of NVP-2203-R1 and NVP-2203-R2)
  Arms: NVP-2203
Drug: NVP-2203-R — administration of active comparator
  Arms: NVP-2203-R

SUMMARY:
The purpose of this study is to evaluate the safety and pharmacokinetics after administration of NVP-2203.

DETAILED DESCRIPTION:
Phase 1 to evaluate the safety and pharmacokinetics after administration of NVP-2203.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult subjects who signed informed consent
* BMI of >18.0 kg/m2 and <30.0 kg/m2 subject, weight more than 50kg(45 kg or more for woman)

Exclusion Criteria:

* Subjects participated in another clinical trial within 6 months prior to administration of the study drug
* Inadequate subject for the clinical trial by the investigator's decision

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2023-05-28 (Actual); Primary Completion 2023-06-11 (Actual); Study Completion 2023-07-05 (Actual)

PRIMARY OUTCOMES:
NVP-2203's pharmacokinetics of plasma | 0hours - 72hours
  AUCt

SECONDARY OUTCOMES:
pharmacokinetics of plasma | 0hours - 72hours
  Cmax

CONTACTS AND LOCATIONS:
Overall Officials: Jaewoo Kim, Principal Investigator — H Plus Yangji Hospital
Locations (1):
- H Plus Yangji Hospital, Seoul, Nambusunhwan-ro, South Korea